CLINICAL TRIAL: NCT05674812
Title: Lung Ultrasound Score Predicts Extubation Failure in Elderly Surgical Patients-- a Multicenterprospective Cohort Study
Brief Title: Extubation Guided by Bedside Ultrasound
Status: Completed | Type: Observational
Sponsor: Lili Jia (Other)
Collaborators: Tianjin Forth Central Hospital (Unknown); Tianjin Fifth Central Hospital (Unknown); Tianjin TEDA Hospital (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Lili Jia, sponsor, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Other Study IDs: TJMZ2022-M001
Record Dates: First submitted 2022-12-08; First posted 2023-01-06 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Insufficiency; Ventilator Weaning; Postoperative Complications
Keywords: Weaning; Ultrasound; Elderly surgical patients
MeSH Terms: conditions — Respiratory Insufficiency; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Extubation Failure: Patients meeting extubation failure criteria within 48 hours after planned extubation
  Interventions: Diagnostic Test: Multimodal pre-extubation risk assessment in elderly surgical patients
- Extubation Success: Patients maintaining spontaneous breathing for >48 hours after extubation
  Interventions: Diagnostic Test: Multimodal pre-extubation risk assessment in elderly surgical patients

INTERVENTIONS:
Diagnostic Test: Multimodal pre-extubation risk assessment in elderly surgical patients — This observational cohort study evaluates risk factors for extubation failure in elderly surgical patients. All participants receive standard pre-extubation clinical assessments per institutional protocol, including LUS、DE and oxygenation index (PaO₂/FiO₂), arterial blood gas analysis, and the patients'laboratory results before and after surgery. The association between these parameters and extubation failure will be analyzed.

SUMMARY:
The aging of the global population has led to an increased number of surgical procedures being performed on elderly patients. However, with aging, the main structure and function of the lungs undergo progressive changes involving lung elasticity , impaired defense mechanisms, weakened respiratory muscle strength, and lessened responsiveness of the lungs to anesthesia . Smetana showed that nearly 33% of patients older than 65 years of age who undergo surgical procedures develop postoperative pulmonary complications. It can be seen that elderly patients are themselves at high risk of pulmonary complications .Common postoperative pulmonary complications include pleural effusion, atelectasis, pneumonia, acute respiratory distress syndrome, cardiogenic pulmonary edema, and postoperative need for mechanical ventilation.This can lead to prolonged hospitalization, increased economic burden on patients, and increased long-term mortality . Therefore, accurately determining factors influencing successful postoperative weaning and extubation in elderly patients is crucial to reduce complications.

Clinical practice guidelines for critically ill patients in general recommend a well-defined, albeit imperfect, protocolized weaning and extubation procedure, including the evaluation of weaning readiness, spontaneous breathing trial (SBT) assessment, extubation, and consideration of prophylactic noninvasive ventilation or high-flow nasal oxygen.However, even if the SBT is successful, 3%-30% of patients still need to be reintubated due to respiratory distress after removal of the endotracheal tube . Predicting successful extubation in these patients is difficult. Predicting successful extubation remains difficult even after a successful SBT. The decision often relies on SBT results and clinical judgment, which can be unreliable. Identifying objective factors associated with extubation failure is therefore essential.

Lung ultrasound score (LUS)has been shown to accurately predict extubation failure by detecting significant pulmonary edema during SBT,and diaphragm excursion (DE)can be used to quantitatively assess diaphragm activity to assess extubation success. However, these studies primarily involved ICU patients with mixed medical and surgical conditions. Data specifically focusing on elderly surgical patients in the Post-Anesthesia Care Unit (PACU) are limited.Given this background, we conducted this multicenter prospective observational study to investigate the association between lung ultrasound parameters (LUS, DE), oxygenation index (OI), and other clinical and laboratory factors with extubation failure specifically in elderly surgical patients recovering in the PACU.

DETAILED DESCRIPTION:
1.1. Research significance mechanical ventilation (MV) is an important technique for the treatment of acute respiratory failure, and about 20% of patients have difficulty in ventilation due to respiratory muscle related diaphragm dysfunction . The duration of mechanical ventilation in elderly patients after large-scale abdominal surgery is longer, the lung function reserve is significantly decreased, and the incidence of postoperative lung complications is as high as 53.1%, which is easy to cause offline difficulties, thus prolongating the hospital stay and seriously threatening the life safety of patients . Therefore, it is of great clinical significance and social value to accurately grasp the ventilator withdrawal time of elderly patients after surgery and reduce ventilator-related lung injury.

1.2. Research status at home and abroad 1.2.1 Research status of mechanical ventilation lung injury Mechanical ventilation provides important respiratory and circulatory support for critically ill patients, but prolonged mechanical ventilation is prone to ventilator-associated lung injury. Studies have shown that with the extension of mechanical ventilation time, the incidence of pulmonary complications increases, such as ventilator-associated pneumonia, which extends the length of ICU stay of patients and increases hospitalization costs . Ventilator-associated diaphragm dysfunction, which has received increasing attention in recent years, is directly related to the duration of mechanical ventilation. Animal studies have shown that the maximum tonic contractile tension and monocontractile tension of diaphragm gradually decrease with the extension of mechanical ventilation . Clinical studies have shown that mechanical ventilation for 18-24 h can lead to diaphragmatic dysfunction . Due to the complicated condition, organ insufficiency and complications of severe patients, it is often very difficult to withdraw the machine. Therefore, the appropriate time of withdrawal is of great significance for the prognosis of elderly critically ill patients.

1.2.2 Characteristics of lung structure and postoperative lung complications in the elderly With the increase of age, the main structure and function of the lung have progressive changes, the lung elastic retraction force is reduced, the defense mechanism is impaired, the respiratory muscle strength is weakened, and the sensitivity to the respiratory depression caused by anesthesia and analgesics is increased, which leads to the decline of the respiratory reserve function. After the trauma stimulation of major surgery for a long time, the lung functional reserve, respiratory muscle strength, lung compliance, respiratory filtration function, gas exchange function and so on decreased significantly in elderly patients. Smetana et al. have shown that the incidence of pulmonary complications in elderly patients after major operations is 33%, the mortality rate of patients within 30 days is 14%30%, the length of hospital stay is prolonged, the medical expenses are increased, and the postoperative quality of life of patients is seriously affected .

Studies have shown that the incidence of postoperative pulmonary complications is negatively correlated with the distance between the surgical site and the diaphragm. The incidence of complications after upper abdominal surgery was 17%76%, and the forced vital capacity after open surgery was reduced by 50% on average, which was positively correlated with the operation duration. Lung complications were 8% if the operation time was less than 2 hours. The complication rate of 34h operation time will increase to 40%. Zuo Mingzhang et al. found that the incidence of pulmonary complications in elderly patients after major abdominal operations was 53.1%. In conclusion, the risk of pulmonary complications after large-scale gastrointestinal abdominal surgery is higher in elderly patients, and the postoperative complications seriously affect the long-term prognosis of patients, prolong the length of hospital stay, and increase hospitalization costs and mortality.

1.2.3 Lung protective ventilation strategies Lung function reserve decreased significantly in elderly patients, and a variety of lung protective ventilation strategies have been applied clinically to reduce the occurrence of postoperative lung complications. Studies have found that the lung protective ventilation strategy of small tidal volume combined with lung reexpansion manipulation can improve lung ventilation function and intrapulmonary oxygenation in elderly patients after major abdominal surgery, reduce postoperative lung complications, and shorten the average length of hospital stay . TAO et al. found that small tidal volume lung ventilation can reduce the occurrence of postoperative lung infection, lung injury and other complications, and to a certain extent reduce the postoperative mortality of patients with general anesthesia . Positive end expiratory pressure (PEEP) reduces the incidence of postoperative atelectasis. Expert consensus on the clinical application of perioperative lung protective ventilation strategy points out that high inhalation oxygen concentration (FiO2) is easy to cause absorptive alveolar collapse and increase the incidence of postoperative lung complications. Helmer horst et al. found that selecting appropriate FiO2 could not only satisfy the oxygen supply of the body and maintain the normal oxygenation index, but also reduce the lung injury caused by high FiO2 .

However, it is of great clinical significance to accurately grasp the timing of extubation, reduce the occurrence of pulmonary complications from the source, and effectively improve the prognosis of elderly patients. Quasha et al. showed that after early extubation, the recovery of respiratory mucosa was accelerated, postoperative pulmonary complications such as atlatasis and pneumonia were significantly reduced, and postoperative outcomes were significantly improved.

At present, the conventional parameters of withdrawal include the following three aspects: (1) Symptom and sign parameters: whether the breathing is coordinated, lung signs, sputum characteristics, patient's consciousness and circulation, etc. (2) Respiratory functional and mechanical parameters: respiratory rate, minute ventilation, vital capacity, airway pressure, lung compliance, etc. (3) Indicators reflecting blood gas exchange: pH, PaO2, PaCO2, etc. In addition, Zhang Xiaofei et al. found that ScvO2 was an early predictor of successful offline extubation in patients with mechanical ventilation, and a decrease of more than 7% in ScvO2 could be used as a prediction threshold. Monitoring ScvO2 was of great significance for the evaluation and management of perioperative critically ill patients, and it could quickly reflect the instantaneous changes in the balance of systemic oxygen supply and demand in critically ill patients. It can detect tissue hypoxia early and is better than other traditional hemodynamic parameters. It is a useful indirect indicator to evaluate whether tissue oxygenation is sufficient or not, and also an important indicator to evaluate the incidence and mortality of perioperative patients with organ failure, infection and other complications. In addition, it was found that arterial oxygen saturation and its change rate had predictive value for the success rate of extubation in patients with mechanical ventilation, and the decrease of SaO2 < 2.6% was a reliable predictor of the success of extubation.

1.2.4 Clinical application status of pulmonary ultrasound

Pulmonary ultrasound, known as a visible stethoscope, can probe the lung condition on the patient's body surface through the ultrasound probe, which can accurately and objectively show the changes of lung ventilation function. The changes of pulmonary ultrasound signs occur earlier than the decline of oxygenation, and have higher sensitivity and accuracy than the traditional chest X-ray. spontaneous breathing test (SBT) is a common clinical off-line extubation test. Spontaneous breathing test (SBT) is a spontaneous extubation test designed to adjust ventilator parameters. PC 5 ~ 8cm H2O, PEEP 5cmH2O, FiO2 < 0.40). At the same time, arterial blood gas was checked once as a reference, and the patient's heart rate, respiration, blood pressure, tidal volume and other parameters, as well as the patient's subjective response (whether dyspnea or not) were recorded every 15min. The results of respiration, circulation, sanity and blood gas were observed within 15min to 2h. Studies have shown that when SBT is used to guide offline, about 15% of patients still fail to take offline and need mechanical ventilation again. Real-time monitoring of lung conditions by lung ultrasound and individualized assessment of lung function and diaphragm function created certain conditions for the early guidance of successful extubation.

Ultrasound assessment of lung function: An increase in the number of lung ultrasound B-lines may reflect the absence of lung ventilation. Therefore, the use of pulmonary ultrasound before and after SBT to evaluate the loss of pulmonary ventilation can predict post-extubation respiratory distress. Soummer et al. used lung ultrasound score (LUS) to quantitatively evaluate lung ventilation. One lung was divided horizontally into upper and lower, and longitudinally into anterior, middle and posterior. The two lungs had 12 regions in total. Scores in each area were evaluated as follows: 0: normal pulmonary ventilation, pulmonary ultrasound showing pulmonary slip sign with A line or less than two isolated B lines; 1 score: moderate lung ventilation loss, lung ultrasound showed 3 or more isolated B lines; 2 points: severe lack of pulmonary ventilation, lung ultrasonography showed combined B-line or curtain sign; 3 points: lung consolidation. LUS varied from 0 to 36 points.

Diaphragmatic dysfunction has a high incidence in severe patients and may lead to a number of pulmonary complications, such as atelectasis and pneumonia. Therefore, early diagnosis of diaphragm dysfunction before extubation can help avoid the risk of extubation failure. Ultrasound can directly observe the left and right diaphragms and how they move with the respiratory cycle. Ji Wenhua et al. examined the degree of diaphragm movement, asked the patient to maintain supine position with the upper abdomen and chest exposed, and after a steady breathing, selected the ultrasonic convex array probe to examine the vertical diaphragm under the costal arch of the bilateral midclavicular line, and the included Angle should be less than 20 °. The M mode was selected to record the distance between the body surface probe and the diaphragm. 30min after SBT, the tracheal catheter was removed, and the distance difference between the expiratory phase and the inspiratory phase was measured after steady breathing, and the movement degree of bilateral diaphragm was detected. The study found that the diaphragm movement degree of the successful extubation group was greater than that of the failed extubation group. At the same time, we also included laboratory indicators before and after surgery to explore the risk factors for extubation failure in elderly surgical patients

ELIGIBILITY:
The inclusion criteria for patients were as follows: aged ≥65 years, underwent general anesthesia for surgery, and were mechanically ventilated for more than 3 hours.

The exclusion criteria for patients were as follows: tracheostomy; inability to perform ultrasound of the diaphragm and parasternal intercostal muscle (morbid obesity, thoracic dressings); central respiratory failure; severe muscle weakness; absence of voluntary diaphragmatic activity; and combined end-stage cardiopulmonary disease; and inability to provide informed consent.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with mechanical ventilation after general anesthesia
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of extubation failure within 48 hours after planned extubation | Within 48 hours after extubation
  Extubation failure was defined as the need for other respiratory support (HFNC, NIV, reintubation) within 48 hours ofplanned extubation.

SECONDARY OUTCOMES:
Mechanical ventilation duration | At the end of the operation, the patient was transferred to the PACU for a short period of ventilatory support, and the last minute of extubation was allowed after awakening and muscle strength recovery
PACU/hospital stay | Patients were observed from the first minute of entering the PACU to the last minute of leaving the PACU/Patients were hospitalized from the first to the last day
postoperative pulmonary complications | Within seven days of surgery
  atelectasis, hypoxemia [SpO2<90% requiring intervention], ARDS, pneumonia, symptomatic pleural effusion, bronchospasm, pneumothorax, aspiration pneumonia
mortality | Mortality within 30 days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Wenli Yu, Principal Investigator — Tian Jin First Center Hospital
Locations (1):
- TianJin First Central Hospital, Tianjin, Tianjin Municipality, China

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT05674812/Prot_ICF_000.pdf